CLINICAL TRIAL: NCT07310342
Title: Physical Fitness of Children, Adolescents and Young Adults With Immune Thrombocytopenic Purpura: a Prospective, Multicentre, Controlled National Study
Brief Title: Physical Fitness of Children, Adolescents and Young Adults With Immune Thrombocytopenic Purpura
Acronym: ITP-CPET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/20; 2025-A00522-47 (Other: ID-RCB number)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Immune thrombocytopenic purpura (ITP); Fatigue; Deconditioning; functional rehabilitation
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Fatigue

STUDY DESIGN:
Intervention Model Description: We aim to compare the cardiopulmonary fitness in children, adolescents, and young adults with chronic ITP to the recently published pediatric reference values [Gavotto, 2023a].
  We plan to express the results for the patient population included in this study in z-scores and by direct comparison with our most recent control group in this study (the most recently published) (n=107).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ITP group (Experimental): Children, adolescents and young adults aged 8 to 25 followed for ITPc (N=53)
  Interventions: Other: IPT-CPET

INTERVENTIONS:
Other: IPT-CPET — Patients with ITP will undergo standard care, medical examination, cardiopulmonary exercise test (CPET), muscular strength and physical activity tests, and validated questionnaires of health-related and disease-related quality of life, mental health, and physical activity

SUMMARY:
Patients with chronic immune thrombocytopenic purpura (ITP) live with an anxiety-inducing risk of haemorrhage that is unpredictable over several months or years.

They also rate fatigue as one of the most frequent (48%) and most severe (73%) disabling symptoms, which contributes to a reduced quality of life [Cooper, 2021].

In this autoimmune disease targeting platelets, fatigue could be mediated by platelet and immunological abnormalities, and/or promoted by psychobehavioural determinants that are poorly understood in this chronic disease.

Since 1980, the World Health Organisation has stated that functional capacity assessments best reflect the impact of chronic diseases on quality of life, with fatigue playing an important role. The association between fatigue and aerobic physical capacity, determined by maximum oxygen consumption (VO2max), has been demonstrated in several pathologies. It is often associated with the vicious circle of deconditioning, where the impact of the disease on cardiac, muscular and respiratory functions is intertwined with inactive or sedentary behaviours.

At the end of this vicious circle, adults have been shown to have an increased cardiovascular risk and a high prevalence of anxiety and depression syndromes.

VO2max measured by cardiopulmonary exercise testing (CPET) is increasingly used in monitoring, as recommended by the French Society of Cardiology [Marcadet, 2018;Marcadet, 2019]. Our team (Amedro et al.) has set up a research programme on aerobic physical capacity and deconditioning to exercise in chronic childhood diseases and has just published the reference values for exercise tests in healthy paediatric populations, enabling the interpretation of VO2max results in sick children [Gavotto,2023].

However, it has been demonstrated that the VO₂ plateau is not predominantly reached in healthy adults and is rarely reached (<25%) in healthy children. [Armstrong, 1996 ; Åstrand, 1952 ; Rowland, 1992].

Thus, the highest oxygen consumption measurement (VO2pic) is often used instead of VO2max to define aerobic capacity. We will therefore use the concepts of VO2max and VO2pic in this study.

The first population studied by our team was children with congenital heart disease, who showed a significant reduction in their VO2max [Amedro, 2018]. Based on these results, a functional rehabilitation programme (QUALIREHAB) was set up and evaluated in a randomised controlled clinical trial [Amedro, 2019] . The data demonstrate its positive impact not only on VO2max, but also on quality of life. Aerobic physical capacity was assessed in chronic paediatric diseases without direct cardiac involvement.

We have also shown that VO2max declines more rapidly over time in children, adolescents and young adults who have survived childhood cancer [Gavotto, 2023] or in children with asthma [Moreau, 2023].

To date, no prospective controlled studies have reported on the level of aerobic physical capacity in children, adolescents and young adults with cITP.

We therefore hypothesise that fatigue in patients monitored for cITP could be correlated with a decrease in their aerobic physical capacity, causing these patients to enter a 'vicious cycle of deconditioning'. If this hypothesis is verified, an exercise rehabilitation programme could have a positive impact on quality of life, physical health and mental health

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents and young adults aged 8 to 25 followed for ITPc
* Patient referred as part of routine care by a CEREVANCE network expert physician to an exercise physiology laboratory for fitness assessment

Exclusion Criteria:

* Presence of at least one contraindication to performing an exercise test

  * Acute anemia < 9g or poorly tolerated chronic anemia, fever, uncontrolled asthma, respiratory failure, acute myocarditis or pericarditis, uncontrolled arrhythmias causing symptoms or hemodynamic disturbance, uncontrolled heart failure, acute pulmonary embolism or pulmonary infarction,
  * Patients with mental impairment leading to an inability to cooperate, as assessed by the physician during the history,
  * Clinical examination abnormalities (heart murmur, rhythm disorders).
* Opposition to participation expressed by the parent(s) or legal guardian(s) for minors (<18 years) or by the patient.
* Absence of social security

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
VO2max measured by exercise testing | Day 1
  Values will be standardised using paediatric reference values.

SECONDARY OUTCOMES:
First ventilatory threshold (SV1) | Day 1
  as a percentage of theoretical VO2max
Ventilatory efficiency | Day 1
  VE/VCO2 slope
Maximal power | Day 1
Oxygen pulse | Day 1
Maximum heart rate | Day 1
Respiratory exchange ratio | Day 1
Respiratory reserve | Day 1
Health-related quality of life | Day 1
  PedsQL®
Disease-specific quality of life | Day 1
  Kids ITP Tools
Muscular force evaluation | Day 1
  Handgrip®
Muscular force evaluation | Day 1
  standing long jump
Physical activity evaluation | Between Day 1 and Day 7
  level of physical activity evaluated using an accelerometer
Physical activity evaluation | Day 1
  * Children and Adolescents Physical Activity and Sedentary Questionnaire
  * International Physical Activity Questionnaire
Mental health evaluation | Day 1
  * Strenghts and difficulties questionnaire
  * Adolescent Depression Rating Scale
  * Patient Health Questionnaire (PHQ-9)
Fatigue evaluation | Day 1
  Fat-PTI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD,PhD, Study Director — University Hospital, Bordeaux; Nathalie ALADJIDI, MD, Study Director — University Hospital, Bordeaux; Marion AUDIE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - Armand de Villeneuve Hospital - Montpellier University Hospital, Montpellier, France
  - Institut Saint-Pierre, Palavas-les-Flots, France
  - Armand Trousseau Hospital - AP-HP, Paris, France
  - Robert Debré Hospital - APHP, Paris, France
  - Pellegrin Hospital - Bordeaux University Hospital, Talence, France